CLINICAL TRIAL: NCT03325231
Title: Factors Influencing Patient Choice of Bladder Reconstruction Following Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: Swansea University (Other)
Collaborators: Abertawe Bro Morgannwg University Health Board (Other)
Responsible Party: Principal Investigator, Prof Phil Reed, Professor, Swansea University
Other Study IDs: RIO 018-17
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder Cancer Patients: Participants will be recruited from those who have had advanced bladder cancer (grade pT1 and above) and undergone either IC or NB procedures within the last five years. No form of payment will be offered for participation, but participants will be reimbursed for travel expenses. There will be no other inclusion or exclusion criteria in order to access a wide range of patients with potentially different values and lifestyles, and to aid in the recruitment of adequate sample sizes.
  Interventions: Other: Reconstructive surgery following bladder removal.

INTERVENTIONS:
Other: Reconstructive surgery following bladder removal. — Investigating patient experience of bladder reconstructions.

SUMMARY:
Radical cystectomy (bladder removal) after bladder cancer necessitates surgical reconstruction to allow urine drainage. Usually, this is achieved by either ileal conduit (a stoma leads to an external bag) or orthotopic neobladder (the creation of an artificial internal bladder). These treatments are most successful when tailored to the patient's own lifestyle needs. The current project will explore patient concerns, and the aspects of their lifestyles and values, that influence their choice of bladder reconstruction. It will also examine which of these concerns and values best predict satisfaction and enhanced QoL, following bladder reconstruction. Participants will be recruited from Health Board databases of those who have had advanced bladder cancer (grade pT1 and above) and undergone either IC or NB procedures within the last five years. 40 participants (equal numbers with each surgical procedure) will be randomly selected from the patient databases. They will be interviewed by a Researcher and a Clinical Nurse Specialist. A semi-structured interview will be conducted to ascertain patients' views about the key factors influencing their treatment decision and their satisfaction with the outcome. Approximately 200 participants (equal numbers with IC and NB) will be sent three questionnaires to assess their life values, QoL, and satisfaction with treatment: (1) Bladder Reconstruction Satisfaction Questionnaire measuring levels of satisfaction with bladder reconstruction; (2) EORTC QLQ-C30 measuring QoL in areas relevant to cancer patients; and (3) Life Values Inventory measuring values and lifestyles important to patients. Participants will be asked to complete the questionnaires and return them using a prepaid envelope. Participants will be provided with the contact details of a Clinical Nurse Specialist known to them to contact if they require help completing the questionnaires.

DETAILED DESCRIPTION:
Aims and Objectives. The proposed research aims: firstly, to enhance our understanding of patient concerns, lifestyles, and values, that influence their choice of bladder reconstruction and predict their treatment satisfaction and quality of life (QoL); and, secondly, to initiate the development a novel decision-aid tool to help bladder-cancer patients, their families, and medical/health professionals to choose the reconstructive surgery following bladder removal that best suits a patient's needs. To these ends, a complementary combination of qualitative and quantitative research approaches will be employed to obtain information from patients about the reasons for their reconstructive surgery choices, the aspects of their lifestyle that were most important to them in reaching their decisions, and the degree to which they are satisfied with their reconstruction. These findings will be used to inform the items to be contained in a pilot joint decision-making tool to support patients and medical professionals when planning such life-changing surgery. Such a tool ultimately could support patient choice, enhance QoL, and influence decision-making practice. Thus, the specific objectives of the research will be to: (1) identify the factors important for patients when choosing a bladder reconstruction; (2) establish the degree to which these factors predict satisfaction with the reconstruction; and, ultimately, (3) start to develop a joint decision-aid tool for patients and medical staff, to use when deciding on the choice of diversionary procedure, that highlights these key factors predicting success and better QoL following different forms of bladder reconstruction.

Methodology and Project Plan. Participants Participants will be recruited from Health Board databases of those who have had advanced bladder cancer (grade pT1 and above) and undergone either IC or NB procedures within the last five years. Around 40 patients per year are referred to the ABMU; this is in line with expectations, given the size of the ABMU patient population (600,000) and rates of bladder cancer, giving a potential sample of 200 patients over the previous five years. This will provide an adequate population from which to sample participants. No form of payment will be offered for participation, but participants will be reimbursed for travel expenses. There will be no other inclusion or exclusion criteria in order to access a wide range of patients with potentially different values and lifestyles, and to aid in the recruitment of adequate sample sizes.

Qualitative Study Forty participants (equal numbers with each surgical procedure) will be randomly selected from the patient databases and invited for interview. This number is achievable given the size of the database, and exceeds the usual criteria (12-18; Guest et al., 2006) for saturation in qualitative research, even with expectation of some non-participation.

The participants will be interviewed by a Researcher and a Clinical Nurse Specialist in a quiet room in the Clinical Research Unit of the Hospital. A semi-structured interview format will be adopted to allow participants latitude in expressing issues that are important to them, and without forcing particular issues. The same semi-structured interview script will be used for each participant, ensuring all are asked the same questions. The general themes to be asked about will be: Who patients consulted and discussed options with; What types of information, support, and advice were they offered; What were the attributes or aspects of the NB/IC that influenced their choice; Which aspects of their lifestyle were most important in making a decision; What factors could have been considered that were not; What types of help have they been offered since; Could they have been offered other information at the time; How do they feel their choice influences their life today; Are they satisfied with their decision. These questions will allow a wide range of patient needs, values, and experiences to be elicited.

Transcribed interview recordings will be subjected to thematic content analysis, in line with previous recommendations (Vaughn et al., 1996), and accepted procedures in health contexts (Osborne et al., 2012a; 2012b; Osborne & Reed, 2008). Transcripts will be examined independently by two Researchers to identify key themes and ensure reliability. Individual 'units of information' contained within each transcript will be highlighted (a 'unit' is any piece of text that relates to an identified theme, and that can be interpreted on its own to provide a meaningful and informative comment). From reading the unitised comments, the initial themes will be refined, so that all 'units of information' can be categorised according to those themes. Coding of 'units' into themes will be conducted independently by two Researchers, and Cohen's Kappa will be used to establish reliability.

Quantitative Study One hundred participants (equal numbers with IC and NB) will be randomly selected from the Health Board database, as described above. The numbers in the database (200) will allow recruitment of these participants, and, assuming a 50% non-return rate, this will allow sufficient power for subsequent analyses. G-Power calculations suggest that, to identify a moderate relationship (r = .3) with 85% power, a sample size of 90 will be needed. If recruitment appears to be low, then other health boards (in particular, Newcastle with whom Mr. Younis is currently employed) will be approached.

Participants will be asked to complete three questionnaires and to return them using a prepaid envelope. Participants will be provided with contact details of a Clinical Nurse Specialist known to them if they require help completing three questionnaires: Bladder Reconstruction Satisfaction Questionnaire measures levels of satisfaction with bladder reconstruction, the relative ease of adapting to the new bladder, and specific aspects patients are happy or unhappy with regarding their procedure; EORTC QLQ-30 (Aaronson et al., 1993) assesses QoL aspects relevant to cancer patients concerning: physical functioning; role functioning; emotional functioning; cognitive functioning; social functioning; and global health status. This questionnaire is reliable and has been used by a large number of researchers (Mystakidou et al., 2001); The Life Values Inventory (Crace & Brown, 1996) measures values across: achievement, belonging, concern for the environment, concern for others, creativity, financial prosperity, health and activity, humility, independence, loyalty to family or group, privacy, responsibility, scientific understanding, and spirituality. The internal reliability is high (Cheng & Fleischmann, 2010).

The values identified will be related by regression analyses to QoL and satisfaction in order to identify whether there are different predictors of outcome for different forms of bladder reconstruction.

Pilot Tool Development Converging themes emerging from the two studies in terms of predicting satisfaction with IC and NB will be drawn together, and a decision-aid tool will be produced for future study. The items identified for inclusion in the tool will be sent to a range of health professionals involved in delivery of surgery and physiotherapy (consultant surgeons, registrars, clinical nurse specialists, and past patients) to obtain their views on its face validity. Items that are rated as inappropriate or redundant will be re-assessed and potentially excluded from the tool, and any missing areas of importance identified by the expert panel will be re-examined.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited from those who have had advanced bladder cancer (grade pT1 and above) and undergone either ileal conduit (IC) or neobladder (NB) procedures within the last five years. There will be no other inclusion criteria in order to access a wide range of patients with potentially different values and lifestyles, and to aid in the recruitment of adequate sample sizes.

Exclusion Criteria:

* Anybody under the age of 18 years will be excluded. Apart from this, there will be no exclusion criteria in order to access a wide range of patients with potentially different values and lifestyles, and to aid in the recruitment of adequate sample sizes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from those who have had advanced bladder cancer (grade pT1 and above) and undergone either ileal conduit (IC) or neobladder (NB) procedures within the last five years.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Bladder Reconstruction Satisfaction Questionnaire | 2 Years
EORTC QLQ-30 | 2 Years
The Life Values Inventory | 2 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Phil Reed, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No